CLINICAL TRIAL: NCT01785615
Title: Interactions of Thrombogenic, Lipogenic, and Inflammatory Markers in Women With the Metabolic Syndrome - Effect of Atorvastatin
Brief Title: Prothrombotic Inflammatory Markers in Women With Metabolic Syndrome - Effect of Atorvastatin
Acronym: PINK
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Gladys Velarde, Principle Investigator, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Protocol No. 1988; Grant# 2004-1035 (Other Grant/Funding Number: RSRB 29937)
Record Dates: First submitted 2013-02-01; First posted 2013-02-07 (Estimated); Results first posted 2017-06-07 (Actual); Last update posted 2017-06-07 (Actual); Status verified 2017-04

CONDITIONS: Metabolic Syndrome
Keywords: metabolic syndrome; atorvastatin; women
MeSH Terms: conditions — Metabolic Syndrome | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorvastatin (Experimental): 44 women randomized to 80 mg atorvastatin for 6weeks
  Interventions: Drug: Atorvastatin
- sugar pill (Placebo Comparator): 44 women randomized to placebo for 6 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Atorvastatin — 80mg
  Other Names: Lipitor
  Arms: Atorvastatin
Other: Placebo — 80mg
  Arms: sugar pill

SUMMARY:
Little is known regarding the association of individual components of the metabolic syndrome (MBS) and prothrombotic, inflammatory and preclinical cardiac structural and functional markers in women with this syndrome. Less is known about adequate treatment as the pathological mechanism of this syndrome is not well understood.

The purpose of this study is two fold;

1. To determine basic differences in biochemical and cardiovascular structural markers in women with and those without MBS and their association with the individual components of MBS.
2. To determine the impact of atorvastatin to lower the risk factors of Metabolic Syndrome. Atorvastatin is one of the most effective drugs approved by the United States Food and Drug Administration (FDA) for the treatment of high cholesterol. It belongs to a class of drugs called statins and its role in primary prevention is still unclear. Thus this population seems to be an ideal group that may benefit from this intervention.

DETAILED DESCRIPTION:
The first phase of the study is an observational phase as previously described. The second phase was a prospective evaluation of the effect of a well known "statin" drug (Lipitor) on different biochemical factors measured in the blood. The eligible study participants had blood work done upon enrollment and if criteria was met(according to the Adult Treatment Panel III), they were given dietary counseling (NYHA - New York Heart Association Step 1 diet) as a lead in phase. Lab work was repeated at 3 weeks to evaluate the impact of the diet and if participant's profile still met criteria for MBS,randomization for either atorvastatin (Lipitor) 80mg or placebo (sugar pill) for 12 weeks took place.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18-75 with Metabolic syndrome
* Abdominal circumference > 35 in
* Hypertriglyceridemia > 150mg/dl
* HDL <50
* Blood Pressure >130/85
* Fasting Glucose >100

Exclusion Criteria:

* Pregnant or planning to become pregnant in the next 6-12 months
* Receiving lipid-lowing drugs
* Obstructive hepatobiliary disease or serious hepatic disease
* Diabetes, cardiovascular disease (CVD), hypothyroidism, active infection, cancer, recent surgery
* Fulfill criteria to receive statin based on LDL levels, risk factors, and Framingham risk scoring outlined on ATP111/NCEP 111 recommendations
* Documented allergic reaction to statin in past
* unexplained elevation in creatinine kinase levels > 3 times upper limit

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2004-11; Primary Completion 2011-12 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gladys P Velarde, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

REFERENCES:
- [Derived] Velarde GP, Choudhary N, Bravo-Jaimes K, Smotherman C, Sherazi S, Kraemer DF. Effect of atorvastatin on lipogenic, inflammatory and thrombogenic markers in women with the metabolic syndrome. Nutr Metab Cardiovasc Dis. 2021 Feb 8;31(2):634-640. doi: 10.1016/j.numecd.2020.10.002. Epub 2020 Oct 10. PMID 33485731

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approximately 250 women volunteers were screened and 140 were selected to go on to the first phase of the trial. After a 6-week period of a run in diet phase, 24 did not return to start randomization. Out of 116 women, 6 failed to meet MBS criteria by one ATP III element.
Groups:
- Atorvastatin: 44 women with metabolic syndrome randomized to 80 mg atorvastatin for 6weeks
  Atorvastatin : 80mg
- Sugar Pill: 44 women with metabolic syndrome randomized to placebo for 6 weeks
  Placebo : 80mg
- Healthy Women: Women without metabolic syndrome
- Metabolic Syndrome Women: These were women who were later randomized to receive Atorvastatin or placebo during phase 2.
Period: Dietary Phase
Arm/Group | Atorvastatin | Sugar Pill | Healthy Women | Metabolic Syndrome Women
Started | 0 | 0 | 35 | 140
Completed | 0 | 0 | 35 | 116
Not Completed | 0 | 0 | 0 | 24
Not completed — Lost to Follow-up | 0 | 0 | 0 | 24
Period: Atorvastatin Phase
Arm/Group | Atorvastatin | Sugar Pill | Healthy Women | Metabolic Syndrome Women
Started | 44 | 44 | 0 | 0
Completed | 44 | 44 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Atorvastatin: 44 women randomized to 80 mg atorvastatin for 6weeks
  Atorvastatin : 80mg
- Sugar Pill: 44 women randomized to placebo for 6 weeks
  Placebo : 80mg
- Total: Total of all reporting groups
Arm/Group | Atorvastatin | Sugar Pill | Healthy Participants | Total
Number analyzed (Participants) | 44 | 44 | 35 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (9) | 52 (9) | 53.7 (9.0) | 52.1 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 44 | 35 | 123
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 44 | 44 | 35 | 88

OUTCOME MEASURES:

1. Primary Outcome: Mean Low Density Lipoprotein Cholesterol in Blood
Description: Approximately 30 ml of blood was collected in two serum (red top), four 3.2% (0.105M) sodium citrate (blue top) Vacutainer® tubes and a syringe at each visit. Collected samples were centrifuged within an hour of collection at 3000xG for 15 minutes at 20°C to obtain platelet-poor plasma and complete serum separation. Each sample was sent to the University of Rochester Clinical Laboratories for testing.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Atorvastatin | Sugar Pill
Number analyzed (Participants) | 44 | 44
mg/dl | 70 (24.8) | 135 (31.4)

2. Primary Outcome: Mean Triglycerides in Blood
Description: as for outcome 1
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Atorvastatin | Sugar Pill
Number analyzed (Participants) | 44 | 44
mg/dl | 139 (54.84) | 185 (65.4)

3. Primary Outcome: Mean Apolipoprotein B in Blood
Description: as for outcome 1
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Atorvastatin | Sugar Pill
Number analyzed (Participants) | 44 | 44
mg/dl | 63 (23) | 110 (23)

4. Primary Outcome: Mean Apolipoprotein B/ Apolipoprotein A1 Ratio in Blood
Description: Approximately 30 ml of blood was collected in two serum (red top), four 3.2% (0.105M) sodium citrate (blue top) Vacutainer® tubes and a syringe at each visit. Collected samples were centrifuged within an hour of collection at 3000xG for 15 minutes at 20°C to obtain platelet-poor plasma and complete serum separation. Each sample was sent to the University of Rochester Clinical Laboratories for testing. The ratio of Apo B to Apo A1 ratio was calculated.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Atorvastatin | Sugar Pill
Number analyzed (Participants) | 44 | 44
ratio | 0.48 (0.18) | 0.86 (0.19)

5. Primary Outcome: Mean High Sensitivity C-reactive Protein in Blood
Description: as for outcome 4
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: ng/dl
Arm/Group | Atorvastatin | Sugar Pill
Number analyzed (Participants) | 44 | 44
ng/dl | 3095 (1778.8) | 4027 (1583.8)

6. Primary Outcome: Mean Waist Circumference
Description: Waist circumference was measured with a ruler tape.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | Atorvastatin | Sugar Pill
Number analyzed (Participants) | 44 | 44
inches | 41.29 (5.13) | 42.79 (4.91)

7. Primary Outcome: Mean Systolic Blood Pressure
Description: Measured with a blood pressure cuff
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Atorvastatin | Sugar Pill
Number analyzed (Participants) | 44 | 44
mm Hg | 130.9 (13.03) | 130.4 (13.30)

8. Primary Outcome: Mean Diastolic Blood Pressure
Description: Measured with a blood pressure cuff
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Atorvastatin | Sugar Pill
Number analyzed (Participants) | 44 | 44
mm Hg | 83.16 (8.67) | 81.86 (8.14)

9. Primary Outcome: Mean High Density Lipoprotein Cholesterol in Blood
Description: as for outcome 1
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Atorvastatin | Sugar Pill
Number analyzed (Participants) | 44 | 44
mg/dl | 46.4 (8.96) | 44.2 (9.35)

10. Primary Outcome: Mean Fasting Plasma Glucose in Blood
Description: as for outcome 1
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Atorvastatin | Sugar Pill
Number analyzed (Participants) | 44 | 44
mg/dl | 90 (25.2) | 93 (16.0)

11. Primary Outcome: Mean Aspartate Aminotransferase in Blood
Description: as for outcome 1
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units/L
Arm/Group | Atorvastatin | Sugar Pill
Number analyzed (Participants) | 44 | 44
units/L | 20.27 (5.73) | 21.09 (7.12)

12. Primary Outcome: Mean Alanine Aminotransferase in Blood
Description: as for outcome 1
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units/L
Arm/Group | Atorvastatin | Sugar Pill
Number analyzed (Participants) | 44 | 44
units/L | 21.59 (9.10) | 23.75 (9.62)

13. Primary Outcome: Mean Leptin in Blood
Description: as for outcome 1
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Atorvastatin | Sugar Pill
Number analyzed (Participants) | 44 | 44
pg/ml | 43077 (24706.7) | 46721.3 (22137.6)

14. Primary Outcome: Mean Soluble Intercellular Adhesion Molecule in Blood
Description: as for outcome 1
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Atorvastatin | Sugar Pill
Number analyzed (Participants) | 44 | 44
ng/ml | 192 (64) | 220 (58)

15. Primary Outcome: Mean Soluble Vascular Adhesion Molecule in Blood
Description: as for outcome 1
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Atorvastatin | Sugar Pill
Number analyzed (Participants) | 44 | 44
ng/ml | 512.9 (121.6) | 534.4 (116.0)

16. Primary Outcome: Mean Plasminogen Activator Inhibitor-1 in Blood
Description: as for outcome 1
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Atorvastatin | Sugar Pill
Number analyzed (Participants) | 44 | 44
ng/ml | 6.18 (0.93) | 6.60 (1.03)

17. Primary Outcome: Mean Myeloperoxidase in Blood
Description: as for outcome 1
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Atorvastatin | Sugar Pill
Number analyzed (Participants) | 44 | 44
ng/ml | 52.18 (16.10) | 59.19 (16.56)

18. Secondary Outcome: Mean Waist Circumference
Description: Waist circumference was measured with a ruler tape.
Time Frame: week 0
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | Healthy Women | Metabolic Syndrome Women
Number analyzed (Participants) | 35 | 88
inches | 33.3 (5.3) | 42.6 (5.7)

19. Secondary Outcome: Mean Low Density Lipoprotein Cholesterol in Blood
Description: as for outcome 1
Time Frame: 0 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- Metabolic Syndrome Women: Women without metabolic syndrome. These were women who were later randomized to receive Atorvastatin or placebo during phase 2.
Arm/Group | Healthy Women | Metabolic Syndrome Women
Number analyzed (Participants) | 35 | 88
mg/dl | 119.9 (24.4) | 133.3 (33.9)

20. Secondary Outcome: Mean Triglycerides in Blood
Description: as for outcome 1
Time Frame: 0 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Healthy Women | Metabolic Syndrome Women
Number analyzed (Participants) | 35 | 88
mg/dl | 94.6 (53.1) | 197.4 (101.6)

21. Secondary Outcome: Mean Myeloperoxidase in Blood
Description: as for outcome 1
Time Frame: 0 weeks
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Healthy Women | Metabolic Syndrome Women
Number analyzed (Participants) | 35 | 88
ng/ml | 43.7 (9.8) | 52.3 (17.1)

22. Secondary Outcome: Mean Fasting Blood Glucose in Blood
Description: as for outcome 1
Time Frame: 0 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Healthy Women | Metabolic Syndrome Women
Number analyzed (Participants) | 35 | 88
mg/dl | 84.3 (11.4) | 95.7 (21.4)

23. Secondary Outcome: Mean High Density Lipoprotein Cholesterol in Blood
Description: as for outcome 1
Time Frame: 0 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Healthy Women | Metabolic Syndrome Women
Number analyzed (Participants) | 35 | 88
mg/dl | 66.6 (9.4) | 46.3 (10.1)

24. Secondary Outcome: Mean Intercellular Adhesion Molecule in Blood
Description: as for outcome 1
Time Frame: 0 weeks
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Healthy Women | Metabolic Syndrome Women
Number analyzed (Participants) | 35 | 88
ng/ml | 179.2 (39.9) | 212.9 (70.2)

25. Secondary Outcome: Mean Systolic Blood Pressure
Description: Measured with a blood pressure cuff
Time Frame: 0 weeks
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Healthy Women | Metabolic Syndrome Women
Number analyzed (Participants) | 35 | 88
mm Hg | 114.5 (12.6) | 132.3 (82.9)

26. Secondary Outcome: Mean Diastolic Blood Pressure
Description: Measured with a blood pressure cuff
Time Frame: 0 weeks
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Healthy Women | Metabolic Syndrome Women
Number analyzed (Participants) | 35 | 88
mm Hg | 74.6 (7.1) | 82.9 (8.3)

27. Secondary Outcome: Mean Vascular Adhesion Molecule in Blood
Description: as for outcome 1
Time Frame: 0 weeks
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Healthy Women | Metabolic Syndrome Women
Number analyzed (Participants) | 35 | 88
ng/ml | 614.8 (108.9) | 525.0 (127.4)

28. Secondary Outcome: Mean Apolipoprotein A-1 in Blood
Description: as for outcome 1
Time Frame: 0 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Healthy Women | Metabolic Syndrome Women
Number analyzed (Participants) | 35 | 88
mg/dl | 172.0 (17.4) | 134.3 (24.0)

29. Secondary Outcome: Mean Apolipoprotein B in Blood
Description: as for outcome 1
Time Frame: 0 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Healthy Women | Metabolic Syndrome Women
Number analyzed (Participants) | 35 | 88
mg/dl | 86.3 (14.9) | 107.2 (23.1)

30. Secondary Outcome: Mean Apolipoprotein B/ Apolipoprotein A1 Ratio in Blood
Description: as for outcome 4
Time Frame: 0 weeks
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Healthy Women | Metabolic Syndrome Women
Number analyzed (Participants) | 35 | 88
ratio | 0.5 (0.1) | 0.8 (0.2)

31. Secondary Outcome: Mean Hs-C Reactive Protein in Blood
Description: as for outcome 1
Time Frame: 0 weeks
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Healthy Women | Metabolic Syndrome Women
Number analyzed (Participants) | 35 | 88
ng/ml | 1761.5 (1520.4) | 3586.9 (1531.7)

32. Secondary Outcome: Mean Leptin in Blood
Description: as for outcome 1
Time Frame: 0 weeks
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Healthy Women | Metabolic Syndrome Women
Number analyzed (Participants) | 35 | 88
pg/ml | 16285.3 (13317.9) | 45518.1 (25798.8)

33. Secondary Outcome: Mean Plasminogen Activator Inhibitor-1 in Blood
Description: as for outcome 1
Time Frame: 0 weeks
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Healthy Women | Metabolic Syndrome Women
Number analyzed (Participants) | 35 | 88
ng/ml | 4.5 (0.7) | 6.2 (1.1)

ADVERSE EVENTS:
Time Frame: LFTs and CPK were obtained at 6 wks, 12 wks, 18 wks by protocol. Urine for microalbuminuria was measured prior to lead-in diet,at 6-week intervals for the first 18 weeks. Renal clearance was measured at randomization and at the end of study.
Description: Randomized subjects received follow-up phone calls to assess for adverse clinical events, side effects (rash, myalgias, muscle aches, etc.), and overall compliance.An emergency contact telephone line was provided for participants to report any concerns or possible drug reactions at any time during the study.
Arm/Group | Atorvastatin | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 0/44 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No